CLINICAL TRIAL: NCT07047456
Title: Prospective Randomized Controlled Phase III Clinical Study on the Impact of Stem Cell Infusion Timing on the Incidence of Acute Graft-versus-host Disease in Patients With Hematologic Malignancies Following Single-unit Umbilical Cord Blood Transplantation
Brief Title: Effect of Stem Cell Infusion Time on aGVHD in Patients With Hematological Malignancies Post UCBT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: infusion time & UCBT
Record Dates: First submitted 2025-06-23; First posted 2025-07-02 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Acute Graft Versus Host Disease
Keywords: Time of umbilical cord blood infusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the early infused group (Active Comparator): infused umbilical cord blood within 8 am and 9 am
  Interventions: Procedure: Time of umbilical cord blood infusion
- the late infused group (Sham Comparator): infused umbilical cord blood within 11:30 am and 12:30 pm
  Interventions: Procedure: Time of umbilical cord blood infusion

INTERVENTIONS:
Procedure: Time of umbilical cord blood infusion — Randomization of patients according to the time of umbilical cord blood infusion

SUMMARY:
To observe the effect of stem cell infusion on the development of acute graft- versus-host disease (aGVHD) in patients with malignant hematologic diseases after single-unit unrelated cord blood transplantation (sUCBT).

DETAILED DESCRIPTION:
Acute graft-versus-host disease (aGVHD) is a major complication and cause of non-relapse mortality following allogeneic hematopoietic stem cell transplantation (allo-HSCT). The human circadian clock utilizes recurring environmental cues such as light exposure and food intake to establish 24-hour rhythmic variations in sleep, hormone secretion, metabolism, body temperature, and immune function. Current clinical strategies for aGVHD prevention primarily focus on pharmacological or immunomodulatory suppression of donor lymphocyte activity, often overlooking the impact of recipient physiological fluctuations on graft outcomes. Our preliminary studies revealed that the timing of stem cell infusion significantly influences the incidence and severity of aGVHD after sUCBT. Given the lack of prospective clinical trial data internationally regarding the effect of infusion timing on aGVHD development post-allo-HSCT, coupled with potential confounding factors in existing retrospective studies and pilot experiments, this study proposes to randomize patients based on umbilical cord blood infusion timing. The investigation will evaluate how infusion time affects aGVHD incidence, other transplantation-related complications, and long-term survival rates in hematologic malignancy patients undergoing sUCBT.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of malignant hematologic disease before transplantation, age, gender and race are not limited;
* Participants were required to have achieved complete remission with negative minimal residual disease (MRD) prior to transplantation;
* Participants who are proposed to receive sUCBT for the first time;
* Eastern Cooperative Oncology Group (ECOG) score 0-2;
* No serious organ failure and active infection;
* Voluntary open randomized controlled study to observe whether the time of stem cell infusion affects the occurrence of aGVHD after transplantation;
* Each subject must sign an informed consent form (ICF) indicating that he/ she understands the purpose and procedures of the study and is willing to participate in the study; in view of the subject's condition, if the participant's own signature is not conducive to the treatment of his/her condition, the ICF will be signed by the legal representative.

Exclusion Criteria:

* Those with severe organ dysfunction or disease, such as severe disease and dysfunction of the heart, liver, kidneys and pancreas;
* Any life-threatening disease, physical condition, or organ system dysfunction that, in the opinion of the investigator, may compromise participant safety and put the results of the study at unnecessary risk; drug-dependent individuals; participants with uncontrolled psychiatric disorders; and individuals with cognitive dysfunction;
* Participants in other clinical studies that may affect aGVHD within 3 months;
* Those whom the investigator considers unsuitable for enrollment (e.g., those who anticipate that patients will not be able to adhere to the examination and treatment due to financial and other issues).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade III to IV aGVHD | 100 days post transplantation
  The primary endpoint of the study will be the development of aGVHD in the first 100 days post-transplant. Acute GVHD was graded according to the Mount Sinai Acute GVHD International Consortium criteria.

SECONDARY OUTCOMES:
The incidence of grade II to IV aGVHD | 100 days post transplantation
  The cumulative incidence of grade II to IV aGVHD in the first 100 days post-transplant. aGVHD was graded according to the Mount Sinai Acute GVHD International Consortium criteria.
The cumulative incidence of neutrophil engraftment at 42 days after transplantation | 42 days post transplantation
  neutrophil engraftment time was defined as the first of three consecutive days during which the neutrophil count was at least 0.5×10^9/L.
The cumulative incidence of platelet engraftment at 60 days after transplantation | 60 days post transplantation
  Platelet engraftment is defined as independence from platelet transfusion for at least 7 days with a platelet count of more than ≥ 20 × 10^9/L.
The cumulative incidence of transplant-related mortality at 360 days after transplantation | 360 days post transplantation
  The cumulative incidence of transplant-related mortality at 360 days after transplantation
The cumulative incidence of relapse at 360 days after transplantation | 360 days post transplantation
  The cumulative incidence of relapse at 360 days after transplantation
The cumulative incidence of overall chronic GVHD at 360 days after transplantation | 360 days post transplantation
  The severity of chronic GVHD was graded according to the 2014 NIH criteria.
The probability of GVHD-free, relapse-free survival(GRFS) | 360 days post transplantation
  The composite endpoint of GRFS was defined as the first events occurring after transplantation among Grade III to IV aGVHD, moderate to severe cGVHD, relapse, or death for any reason.
The probability of disease-free survival(DFS) | 360 days post transplantation
  The DFS was defined as the interval between transplantation and disease recurrence, death or the last follow-up date, whichever occurred first.
The probability of overall survival(OS) | 360 days post transplantation
  The OS was determined to be the time from the first day of transplantation until death from any cause or the last follow-up date.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyu Zhu, Ph.D, Principal Investigator — The First Affiliated Hospital of USTC
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No